CLINICAL TRIAL: NCT05644184
Title: A Phase 2, Randomized, Observer-blind, Controlled, Age De-escalation, Dosage Escalation Study to Assess Safety and Immunogenicity of a Novel Live Attenuated Type 1 Oral Poliomyelitis Vaccine in Healthy Young Children, Infants, and Neonates in Bangladesh
Brief Title: Study of a Novel Type 1 Oral Poliomyelitis Vaccine in Bangladesh
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); PT Bio Farma (Industry); Centers for Disease Control and Prevention (U.S. Federal Agency); DiagnoSearch Life Sciences Pvt. Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CVIA 093
Record Dates: First submitted 2022-11-10; First posted 2022-12-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Poliomyelitis
Keywords: Vaccine tolerability; Vaccine safety; Vaccine reactogenicity; Vaccine viral shedding; Vaccine immunogenicity
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Intervention Model Description: A 15-arm, randomized, observer-blind, controlled, age de-escalation, dosage escalation study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (15):
- Group 1: Young Children, nOPV1 10^5.5 CCID50 (Experimental): 48 young children aged 1 to <5 years will receive 2 doses of nOPV1 at a dose level of 10^5.5 CCID50 on Day 1 and Day 29
  Interventions: Biological: Novel Live Attenuated Type 1 Oral Poliomyelitis Vaccine (nOPV1)
- Group 3: Young Children, nOPV1 10^6.0 CCID50 (Experimental): 48 young children aged 1 to <5 years will receive 2 doses of nOPV1 at a dose level of 10^6.0 CCID50 on Day 1 and Day 29
  Interventions: Biological: Novel Live Attenuated Type 1 Oral Poliomyelitis Vaccine (nOPV1)
- Group 5: Young Children, nOPV1 10^6.5 CCID50 (Experimental): 48 young children aged 1 to <5 years will receive 2 doses of nOPV1 at a dose level of 10^6.5 CCID50 on Day 1 and Day 29
  Interventions: Biological: Novel Live Attenuated Type 1 Oral Poliomyelitis Vaccine (nOPV1)
- Groups 2, 4 and 6: Young Children, mOPV1 (Active Comparator): 48 young children aged 1 to <5 years will receive 2 doses of mOPV1 at a dose level of ≥ 10^6.0 CCID50 on Day 1 and Day 29
  Interventions: Biological: Sabin Monovalent Oral Poliomyelitis Vaccine Type 1 (mOPV1)
- Group 7: Infants, nOPV1 10^5.5 CCID50 (Experimental): 96 infants aged 6 weeks (+6 days) will receive 1 dose of IPV on Day 1, then 2 doses of nOPV1 at a dose level of 10^5.5 CCID50 on Day 29 and Day 57, and a challenge dose of mOPV on Day 113.
  Interventions: Biological: Novel Live Attenuated Type 1 Oral Poliomyelitis Vaccine (nOPV1); Biological: Sabin Monovalent Oral Poliomyelitis Vaccine Type 1 (mOPV1)
- Group 9: Infants, nOPV1 10^6.0 CCID50 (Experimental): 96 infants aged 6 weeks (+6 days) will receive 1 dose of IPV on Day 1, then 2 doses of nOPV1 at a dose level of 10^6.0 CCID50 on Day 29 and Day 57, and a challenge dose of mOPV on Day 113.
  Interventions: Biological: Novel Live Attenuated Type 1 Oral Poliomyelitis Vaccine (nOPV1); Biological: Sabin Monovalent Oral Poliomyelitis Vaccine Type 1 (mOPV1)
- Group 11: Infants, nOPV1 10^6.5 CCID50 (Experimental): 48 infants aged 6 weeks (+6 days) will receive 1 dose of IPV on Day 1, then 2 doses of nOPV1 at a dose level of 10^6.5 CCID50 on Day 29 and Day 57, and a challenge dose of mOPV on Day 113.
  Interventions: Biological: Novel Live Attenuated Type 1 Oral Poliomyelitis Vaccine (nOPV1); Biological: Sabin Monovalent Oral Poliomyelitis Vaccine Type 1 (mOPV1)
- Group 11b: Infants, nOPV1 10^6.5 CCID50 (Experimental): 96 infants aged 6 weeks (+6 days) will receive 1 dose of IPV on Day 1, then 3 doses of nOPV1 at a dose level of 10^6.5 CCID50 on Day 29, Day 57 and Day 85, and a challenge dose of mOPV on Day 141.
  Interventions: Biological: Novel Live Attenuated Type 1 Oral Poliomyelitis Vaccine (nOPV1); Biological: Sabin Monovalent Oral Poliomyelitis Vaccine Type 1 (mOPV1)
- Group 13: Infants, nOPV1 10^7.0 CCID50 (Experimental): 96 infants aged 6 weeks (+6 days) will receive 1 dose of IPV on Day 1, then 3 doses of nOPV1 at a dose level of 10^7.0 CCID50 on Day 29, Day 57 and Day 85, and a challenge dose of mOPV on Day 141.
  Interventions: Biological: Novel Live Attenuated Type 1 Oral Poliomyelitis Vaccine (nOPV1); Biological: Sabin Monovalent Oral Poliomyelitis Vaccine Type 1 (mOPV1)
- Group 15: Infants, nOPV1 10^7.5 CCID50 (Experimental): 96 infants aged 6 weeks (+6 days) will receive 1 dose of IPV on Day 1, then 3 doses of nOPV1 at a dose level of 10^7.5 CCID50 on Day 29, Day 57 and Day 85, and a challenge dose of mOPV on Day 141.
  Interventions: Biological: Novel Live Attenuated Type 1 Oral Poliomyelitis Vaccine (nOPV1); Biological: Sabin Monovalent Oral Poliomyelitis Vaccine Type 1 (mOPV1)
- Groups 8, 10, 12, 12b, 14, 16: Infants mOPV1 (Active Comparator): 192 infants aged 6 weeks (+6 days) will receive 1 dose of IPV on Day 1 then 2 to 3 doses of mOPV1 at a dose level of ≥10^6.0 CCID50 on Day 29, Day 57, Day 85 (groups 12b, 14 & 16 only) and a challenge dose of mOPV on Day 113 (groups 8, 10 & 12) on Day 141 (groups 12b, 14 & 16)
  Interventions: Biological: Novel Live Attenuated Type 1 Oral Poliomyelitis Vaccine (nOPV1); Biological: Sabin Monovalent Oral Poliomyelitis Vaccine Type 1 (mOPV1)
- Group 17: Neonates, nOPV1 10^6.5 CCID50 (Experimental): 330 neonates (day of birth +3 days) will receive 3 doses of nOPV1 at a dose level of 10^6.5 CCID50 on Day 1, Day 29 & Day 57
  Interventions: Biological: Novel Live Attenuated Type 1 Oral Poliomyelitis Vaccine (nOPV1)
- Group 19: Neonates, nOPV1 10^7.0 CCID50 (Experimental): 330 neonates (day of birth +3 days) will receive 3 doses of nOPV1 at a dose level of 10^7.0 CCID50 on Day 1, Day 29 & Day 57
  Interventions: Biological: Novel Live Attenuated Type 1 Oral Poliomyelitis Vaccine (nOPV1)
- Group 21: Neonates, nOPV1 10^7.5 CCID50 (Experimental): 330 neonates (day of birth +3 days) will receive 3 doses of nOPV1 at a dose level of 10^7.5 CCID50 on Day 1, Day 29 & Day 57
  Interventions: Biological: Novel Live Attenuated Type 1 Oral Poliomyelitis Vaccine (nOPV1)
- Groups 18, 20 & 22: Neonates, mOPV1 (Active Comparator): 330 neonates (day of birth +3 days) will receive 3 doses of mOPV1 at a dose level of ≥ 10^6.0 CCID50 on Day 1, Day 29 & Day 57
  Interventions: Biological: Sabin Monovalent Oral Poliomyelitis Vaccine Type 1 (mOPV1)

INTERVENTIONS:
Biological: Novel Live Attenuated Type 1 Oral Poliomyelitis Vaccine (nOPV1) — Drop counts of nOPV vaccine will be varied to achieve approximately 10^5.5, 10^6.0, 10^6.5 CCID50 or 10^7.0, 10^7.5 dose levels.
  Arms: Group 11: Infants, nOPV1 10^6.5 CCID50; Group 11b: Infants, nOPV1 10^6.5 CCID50; Group 13: Infants, nOPV1 10^7.0 CCID50; Group 15: Infants, nOPV1 10^7.5 CCID50; Group 17: Neonates, nOPV1 10^6.5 CCID50; Group 19: Neonates, nOPV1 10^7.0 CCID50; Group 1: Young Children, nOPV1 10^5.5 CCID50; Group 21: Neonates, nOPV1 10^7.5 CCID50; Group 3: Young Children, nOPV1 10^6.0 CCID50; Group 5: Young Children, nOPV1 10^6.5 CCID50; Group 7: Infants, nOPV1 10^5.5 CCID50; Group 9: Infants, nOPV1 10^6.0 CCID50; Groups 8, 10, 12, 12b, 14, 16: Infants mOPV1
Biological: Sabin Monovalent Oral Poliomyelitis Vaccine Type 1 (mOPV1) — The Sabin Monovalent Oral Poliomyelitis Vaccine Type 1 control and challenge vaccine (mOPV1) contains ≥ 10^6.0 CCID50 per 0.1 mL (2 drops) dose.
  Arms: Group 11: Infants, nOPV1 10^6.5 CCID50; Group 11b: Infants, nOPV1 10^6.5 CCID50; Group 13: Infants, nOPV1 10^7.0 CCID50; Group 15: Infants, nOPV1 10^7.5 CCID50; Group 7: Infants, nOPV1 10^5.5 CCID50; Group 9: Infants, nOPV1 10^6.0 CCID50; Groups 18, 20 & 22: Neonates, mOPV1; Groups 2, 4 and 6: Young Children, mOPV1; Groups 8, 10, 12, 12b, 14, 16: Infants mOPV1

SUMMARY:
The purpose of this clinical trial is to assess the safety and tolerability (primary objective), immunogenicity (primary and secondary objectives), fecal shedding of vaccine viruses (secondary objective) and the potential for neurovirulence of shed virus (secondary objective) of a novel oral polio type 1 vaccine, nOPV1, as compared to Sabin monovalent type 1 vaccine controls (mOPV1), in healthy young children (192 subjects), infants (720 subjects), and neonates (1320 subjects).

DETAILED DESCRIPTION:
This single-center trial is the first clinical assessment of nOPV1 in a pediatric population. It will be a 15-arm, randomized, observer-blind, controlled trial, with Sabin monovalent type 1 vaccine (mOPV1) serving as the control. Enrollment in this pediatric study will be staggered into three age-descending cohorts, Cohort 1 composed of 192 healthy young children 1 to less than 5 years of age who have completed their full routine polio immunization series, Cohort 2 composed of 720 healthy infants 6 weeks of age (+6 days) who will receive only one dose of inactivated poliomyelitis vaccine (IPV) on Day 1, and finally Cohort 3, composed of 1320 healthy poliomyelitis unvaccinated neonates (day of birth +3 days). Participants will receive two or three doses of either nOPV1 at dose levels of 10^5.5 CCID50, 10^6.0 CCID50, 10^6.5 CCID50, 10^7.0 CCID50 or 10^7.5 CCID50 or the mOPV control vaccine. The second and third doses of vaccine will be given 28 days following the prior dose. In order to demonstrate the vaccine's ability to reduce fecal shedding following a challenge with the Sabin type 1 strain, the infant cohort will be challenged with mOPV 8 weeks after their last dose of nOPV. Participants will be followed until 28 weeks (young children and neonates) or 32 weeks (infants) after their Day 1 vaccination.

ELIGIBILITY:
Inclusion Criteria for all participants:

1. Healthy, as defined by the absence of any clinically significant medical condition or congenital anomaly as determined by medical history, physical examination, and clinical assessment of the investigator
2. Parent(s) or guardian(s) willing and able to provide written informed consent prior to performance of any study-specific procedure
3. Resides in study area and parent understands and is able and willing to adhere to all study visits and procedures (as evidenced by a signed informed consent form [ICF] and assessment by the investigator)
4. Parent agrees for participant to receive all routine infant and childhood immunizations as per the approved protocol-adjusted schedule

Inclusion Criteria for Cohort 1 (young children) participants only:

1. Male or female child from 1 to less than 5 years of age at the time of initial study vaccination
2. Based on documentation, previously received a 3 or 4 dose primary poliomyelitis immunization series containing OPV (may have also received IPV), with last dose received more than 3 months prior to initial study vaccination

Inclusion Criteria for Cohort 2 (infants) participants only:

1. Male or female infant expected to be 6 weeks of age (43rd to 49th day of life [with day of birth being the first day of life], inclusive+ 6-day window), at the time of initial study vaccination
2. Prior to study vaccination has received no doses of IPV or OPV, based on no evidence of such vaccination per available documentation.

Inclusion Criteria for Cohort 3 (neonates) participants only:

1. Male or female newborn (1st day of life+ 3-day window, inclusive), at the time of initial study vaccination
2. Prior to study vaccination has received no doses of IPV or OPV or rotavirus vaccine, based on no evidence of such vaccination per available documentation.

Exclusion Criteria for all participants:

1. For all participants, the presence of anyone under 10 years of age in the participant's household (living in the same house or apartment unit) who does not have complete "age appropriate" vaccination status with respect to poliovirus vaccines at the time of study vaccine administration. For household members younger than 10 years of age, "age appropriate" vaccination is complete series of trivalent Oral Poliovirus Vaccine (tOPV) or at least three doses of bivalent (types 1 and 3) Oral Poliovirus Vaccine (bOPV) plus a booster fractional dose of IPV (fractional dose Inactivated Polio Vaccine; fIPV). Note: A vaccination series of tOPV or at least three doses of bOPV with our without a booster fractional dose of IPV will be considered sufficient.
2. For all participants, having a member of the participant's household (living in the same house or apartment unit) who has received OPV based on the vaccination records in the previous 3 months before study vaccine administration.
3. Any participating children attending day care or pre-school during their participation in the study until one month after their last study vaccine administration.
4. Moderate or severe (grade ≥ 2) acute illness at the time of enrollment/first study vaccination - temporary exclusion. Participant with mild (grade 1) acute illnesses may be enrolled at the discretion of the investigator.
5. Presence of fever on the day of enrollment/first study vaccination (axillary temperature ≥37.5˚C) - (Temporary exclusion for Cohorts 1 and 2)
6. A known allergy, hypersensitivity, or intolerance to any components of the study vaccines, including all macrolide and aminoglycoside antibiotics (e.g., erythromycin and kanamycin)
7. Evidence of a clinically significant congenital or genetic defect as judged by the investigator
8. History of chronic administration (defined as more than 14 days) of immunosuppressant medications, including corticosteroids (> 0.5mg/kg/day of prednisolone (or equivalent)). Topical and inhaler steroids are permitted (unless indicative of a significant chronic illness otherwise excluding the infant/young child)
9. Any self-reported known or suspected immunosuppressive or immunodeficiency condition (including HIV infection) in the participant or household member (living under the same roof/in the same building rather than in the same compound)
10. Receipt of any immune-modifying or immunosuppressant drugs within 6 months prior to the first study vaccine dose or planned use during the study of study participants or a household member
11. Any known or suspected bleeding disorder in the participant that would pose a risk to venipuncture or intramuscular injection
12. Presence of sever malnutrition [weight-for-length/height z-score greater than or equal to -3 SD median (per WHO published growth standards)] - temporary exclusion if marginal and subsequently gains weight.
13. Participation in another investigational product (drug or vaccine) clinical trial within 30 days prior to entry in this study or receipt of any such investigational product other than the study vaccine within 30 days prior tot he first administration of study vaccine, or planned use during the study period.
14. Receipt of transfusion of any blood product or immunoglobulins within 12 months prior to the first administration of study vaccine or planned use during the study period.
15. Parent or participant has any condition that in the opinion of the investigator would increase the participant's health risks in the study participation or would increase the risk of not achieving the study's objectives (e.g., would compromise adherence to protocol requirements or interfere with planned safety and immunogenicity assessments.)

Exclusion Criteria for Cohort 2 & 3 participants only:

1. Low birth weight (LBW) in newborn participants which is defined as a birth weight of less than 2500g (up to and including 2499b) at the time of birth or by the time of enrolment.
2. Premature birth (less than 37 weeks gestation)
3. From multiple birth (due to increased risk of OPV transmission between siblings)

Ages: 0 Days to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2232 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Frequency of serious adverse events (SAEs) from the time of first study vaccination through the end of the study | From Day 1 to end of study, up to Day 197 (young children and neonates) or Day 225 (infants)
  Serious adverse event is any adverse event that results in any of the following outcomes:
  1. Death
  2. Is life-threatening (life-threatening means that the study participant was, in the opinion of the site PI or PATH, at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe).
  3. Requires inpatient hospitalization or prolongation of existing hospitalization
  4. Results in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
  5. Important medical event that may not result in one of the above outcomes but may jeopardize the health of the study participant and require medical or surgical intervention to prevent one of the outcomes listed in the above definition of serious adverse event
Frequency of solicited adverse events (AEs) for 7 days (day of vaccination and 6 following days) after each vaccination | From vaccination to 7 days post vaccination
  Solicited AEs are pre-specific AEs that are common or known to be associated with vaccination that are actively monitored as potential indicators of vaccine reactogenicity. The following specific solicited AEs will be monitored for this trial:
  * Fever (axillary temperature ≥ 37.5°C)
  * Vomiting
  * Diarrhea
  * Irritability
  * Decreased feeding or appetite
  * Fatigue or decreased activity
Frequency of unsolicited AEs for 28 days (day of vaccination and 27 following days) after each vaccination | From vaccination to 28 days post vaccination
  Unsolicited AEs are any AEs reported spontaneously by the participant's parent, observed by the study personnel during study visits or identified during review of medical records or source documents. In the absence of a diagnosis, abnormal physical examination findings or abnormal clinical safety laboratory test results that are assessed by the investigator to be clinically significant will be reported as an AE.
Post-vaccination frequency of seroconversion of type 1 anti-polio serum neutralizing antibody (NAb). | 28 days post second vaccination
  Following two doses of nOPV1, at dose levels of 10^6.5 and 10^7.0 CCID50/dose, compared to mOPV1, in healthy neonates.
  For unvaccinated neonates, seroconversion will be defined as either a minimum 4-fold higher antibody titer relative to the expected level of maternal antibody and seropositivity (reciprocal titer ≥ 8) at the post-vaccination time point among those initially seropositive, or post-vaccination seropositivity among those initially seronegative.

SECONDARY OUTCOMES:
Post-vaccination frequency of seroconversion of type 1 anti-polio serum NAb. | Baseline and 28 days post vaccination (Day 1 and Day 29 for young children, Day 1, Day 29 and Day 57 for neonates and Day 29, Day 57 and Day 85 for infants)
  To assess the seroconversion rate elicited by nOPV1 at dose levels of 10^6.5, 10^7.0 and 10^7.5 CCID50/dose following one and three doses in healthy neonates compared to mOPV1.
  To assess the seroconversion rate elicited by nOPV1 at dose levels of 10^5.5, 10^6.0 and 10^6.5 CCID50/dose following one or two doses in healthy young children compared to mOPV1.
  To assess the seroconversion rate elicited by nOPV1 at dose levels of 10^5.5 and 10^6.0 CCID50/dose following one or two doses in healthy infants compared to mOPV1.
Median type 1 anti-polio serum NAb titers. | Baseline and 28 days post vaccination (Day 1 and Day 29 for young children, Day 1, Day 29 and Day 57 for neonates and Day 29, Day 57 and Day 85 for infants)
  Elicited by nOPV1, compared to that of mOPV1, following one or two doses in healthy young children, and one, two or three doses in infants and neonates.
Type 1 anti-polio serum NAb Geometric Mean Titer (GMT). | Baseline and 28 days post vaccination (Day 1 and Day 29 for young children, Day 1, Day 29 and Day 57 for neonates and Day 29, Day 57 and Day 85 for infants)
  Elicited by nOPV1, compared to that of mOPV1, following one or two doses in healthy young children, and one, two or three doses in infants and neonates.
Post-vaccination GMT ratios of type 1 anti-polio serum NAb, adjusted for baseline immunity. | Baseline and 28 days post vaccination (Day 1 and Day 29 for young children, Day 1, Day 29 and Day 57 for neonates and Day 29, Day 57 and Day 85 for infants)
  Elicited by nOPV1, compared to that of mOPV1, following one or two doses in healthy young children, and one, two or three doses in infants and neonates.
Seroprotection rate, defined as type 1 anti-polio serum NAb reciprocal titer ≥ 8. | Baseline and 28 days post vaccination (Day 1 and Day 29 for young children, Day 1, Day 29 and Day 57 for neonates and Day 29, Day 57 and Day 85 for infants)
  Elicited by nOPV1, compared to that of mOPV1, following one or two doses in healthy young children, and one, two or three doses in infants and neonates.
Geometric mean fold rise (GMFR) in NAb titer relative to baseline | Baseline and 28 days post vaccination (Day 1 and Day 29 for young children, Day 1, Day 29 and Day 57 for neonates and Day 29, Day 57 and Day 85 for infants)
  Elicited by nOPV1, compared to that of mOPV1, following one or two doses in healthy young children, and one, two or three doses in infants and neonates.
Proportion of participants shedding type 1 poliovirus at any and at each post-vaccination stool collection, as assessed by polymerase chain reaction (PCR) in infants and neonates. | Baseline through to 28 days post initial vaccination (Day 29 through to Day 57 for infants; Day 1 through to Day 29 for neonates)
  28 days after the initial dose of nOPV1, compared to mOPV1.
Proportion of participants shedding type 1 poliovirus at any and at each post-challenge stool collection, as assessed by PCR in infants. | Day of challenge through to 28 days post challenge (Day 113 through to Day 141 or 169, for infants)
  28 days after mOPV challenge compared to mOPV1
Neurovirulence of shed study vaccine virus from select stool samples as measured by a transgenic mouse neurovirulence test in a subset of infants. | Baseline through to 28 days post initial vaccination (Day 29 through 57 for infants)
  Within 28 days of an initial nOPV dose and compared to that of mOPV1.

CONTACTS AND LOCATIONS:
Overall Officials: K. Zaman, MBBS, MPH, PhD, FRCP, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b), Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No